CLINICAL TRIAL: NCT02904603
Title: Prospective Monitoring of Immune Parameters in Patients With Hepatitis C Under Treatment With Direct Acting Antivirals
Brief Title: Immune Monitoring of Hepatitis C Under DAA Therapy
Acronym: IMHC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Dr. Georg Peschel, Dr. med., University of Regensburg
Other Study IDs: IM-HC-1516
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum probes
Oversight: Data Monitoring Committee: No

SUMMARY:
Direct acting antivirals offer a new opportunity to monitor the immune response in Hepatitis C infection. In this study cytokine markers will be measured during therapy up to time point SVR 12 an correlated to clinical Parameters and regular laboratory findings.

ELIGIBILITY:
Inclusion Criteria:

* written consent, age, HCV-RNA positive, DAA therapy

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under DAA therapy > 18 years monocentral.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change of IP10 and related cytokines during treatment (ng/ml) | 24 weeks (observation time under and after DAA therapy)
  Screening for Biomarkers under DAA Therapy until timepoint SVR 12 (12 weeks treatment plus control 12 weeks after end of Treatment = 24 weeks)

SECONDARY OUTCOMES:
SVR 12 | 24 weeks (12 weeks treatment plus control 12 weeks after end of treatment)
  Eradication of HCV RNA 12 weeks after end of Treatment (Treatment 12 weeks)
Change of inflammatory markers (ferritin ng/ml, CRP mg/l, PCT ng/ml) during treatment | 24 weeks (observation time under DAA therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Kilian Weigand, Study Chair — Uiversity of Regensburg
Locations (1):
- University of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adenugba A, Hornung M, Weigand K, Peschel G, Junger H, Kupke P, Lang H, Marquardt JU, Zimmermann T, Geissler EK, Schlitt HJ, Werner JM. Ribavirin Improves NK Cell IFNgamma Response During Sofosbuvir-based DAA Therapy in HCV-infected Liver Transplant Recipients. Transplantation. 2021 Oct 1;105(10):2226-2238. doi: 10.1097/TP.0000000000003612. PMID 33587435
- [Derived] Hutchinson JA, Weigand K, Adenugba A, Kronenberg K, Haarer J, Zeman F, Riquelme P, Hornung M, Ahrens N, Schlitt HJ, Geissler EK, Werner JM. Predicting Early Viral Control under Direct-Acting Antiviral Therapy for Chronic Hepatitis C Virus Using Pretreatment Immunological Markers. Front Immunol. 2018 Feb 7;9:146. doi: 10.3389/fimmu.2018.00146. eCollection 2018. PMID 29467758